CLINICAL TRIAL: NCT07200427
Title: Multimodal Engagement and Sustainable Lifestyle Interventions Optimizing Breast Cancer Risk Reduction Supported by Artificial Intelligence
Brief Title: MELIORA Virtual Coach Intervention for Breast Cancer Prevention
Acronym: MELIORA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: BROSTCANCERFORENINGEN AMAZONA I STOCKHOLMS LAN (Unknown); Karolinska Institutet (Other); Instituto de Investigacion Sanitaria INCLIVA (Other); FUNDACION PARA LA INVESTIGACION DEL HOSPITAL CLINICO DE LA COMUNITAT VALENCIANA, FUNDACION INCLIVA (Unknown); LIETUVOS SVEIKATOS MOKSLU UNIVERSITETAS (Unknown); PAGALBOS ONKOLOGINIAMS LIGONIAMS ASOCIACIJA (Unknown); SWPS UNIWERSYTET HUMANISTYCZNOSPOLECZNY (Unknown); EUROPEAN FOOD INFORMATION COUNCIL (Unknown); PREDICTBY RESEARCH AND CONSULTING S.L. (Unknown); ETHNIKO KENTRO EREVNAS KAI TECHNOLOGIKIS ANAPTYXIS (Unknown); EXUS SOFTWARE MONOPROSOPI ETAIRIA PERIORISMENIS EVTHINIS (Unknown); RISA SICHERHEITSANALYSEN GMBH (Unknown); BIOASSIST SA (Unknown); EUROPEAN HEALTH MANAGEMENT ASSOCIATION (Unknown); ETICAS DATA SOCIETY (Unknown)
Responsible Party: Principal Investigator, Yannis Manios, Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101136791
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Prevention
Keywords: Behavior change; Disease prevention; Health behaviour; Primary prevention; Public and environmental health; Breast cancer; Cancer prevention; Sustainable intervention; Nutrition; Diet; Physical activity; Exercise; Lifestyle; Public health; Cancer risk factors; Health communication; Digital health; Health technologies; Artificial intelligence; randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The MELIORA RCTs will employ a parallel-group, randomized controlled design with two groups: an intervention group and a control group. The study follows a superiority design, with individual-level randomization and a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MELIORA Virtual Coach Intervention (VCI) Group (Experimental): The intervention group will receive generic advice on a healthy lifestyle and breast cancer (BC) prevention plus access to the full MELIORA VCI app.
  Interventions: Behavioral: MELIORA Virtual Coach Intervention
- Control Group (Placebo Comparator): The control group will receive the standard of care that is generic advice for a healthy lifestyle and BC prevention.
  Interventions: Other: Control (generic advice)

INTERVENTIONS:
Behavioral: MELIORA Virtual Coach Intervention — Based on baseline assessments, the MELIORA VCI app will prompt intervention group participants to set weekly goals on lifestyle behaviours such as physical activity, diet, alcohol use, and sedentary time, and support daily self-monitoring and step count tracking. Goals will be dynamically adjusted by the virtual coach or the participant to remain realistic and achievable. Τhe app will also offer culturally adapted educational, motivational, and instructional support through mini-courses, tips, recommendations and an embedded library of relevant materials to ensure high adoption rates among women from diverse countries, socioeconomic backgrounds and minority groups. To boost motivation, it will include reminders, gamification features like badges and points, as well as personalized techniques such as action planning, problem solving, social reward, and positive self-talk.
  Arms: MELIORA Virtual Coach Intervention (VCI) Group
Other: Control (generic advice) — The control group will receive the standard of care that is generic advice for a healthy lifestyle and BC prevention. A 'light' version of the MELIORA VCI app will be developed to host the control group materials, track participants' step counts, send reminders, and allow scheduling of follow-up visits. No other features will be available in this version of the app.
  Arms: Control Group

SUMMARY:
Breast cancer (BC) is the most commonly diagnosed cancer in women worldwide, with early-onset cases increasing due to genetic and lifestyle factors. Traditional prevention strategies have shown limited effectiveness, creating the need for innovative approaches. The MELIORA project develops an AI-driven digital tool, the Virtual Coach (VC), to promote sustainable behaviour change in physical activity, diet, and alcohol use. Three randomized-controlled studies will be conducted: MELIORA-HEALTHY (women at risk, n=1080 in Greece, Lithuania, Spain), MELIORA-PATIENTS (women undergoing treatment, n=400 in Lithuania, Spain), and MELIORA-SURVIVORS (post-treatment survivors, n=600 in Lithuania, Spain, Sweden). Participants across diverse regions and backgrounds will be randomized to standard lifestyle advice or the same advice plus the MELIORA VC app. Each study lasts 12 months, with outcomes assessed at baseline, 6, and 12 months. The primary outcome is physical activity, with secondary outcomes including sedentary behaviour, diet, alcohol use, and quality of life. If effective, the MELIORA VC could offer a scalable, cost-effective model for BC prevention and survivorship care, providing valuable evidence to guide public health strategies.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most commonly diagnosed cancer among women worldwide, with early-onset cases rising rapidly due to interactions between genetics and lifestyle behaviours. Traditional efforts to modify these behaviours have had limited success, highlighting the need for innovative, multifaceted approaches. The Multimodal Engagement and Sustainable Lifestyle Interventions Optimizing Breast Cancer Risk Reduction Supported by Artificial Intelligence (MELIORA) project addresses this gap by promoting sustainable behaviour change through an innovative intervention using artificial intelligence (AI). The project will develop and evaluate an AI-driven behaviour change digital solution, the MELIORA virtual coach (VC), designed to enhance awareness, motivation, and promote healthier lifestyle choices related to physical activity, diet, and alcohol consumption, while addressing potential implementation barriers.

The MELIORA VC intervention consists of three separate studies: 1) the MELIORA-HEALTHY Study targeting healthy women at risk of BC (conducted in Greece, Lithuania, Spain), 2) the MELIORA-PATIENTS Study targeting BC patients (conducted in Lithuania, Spain), and 3) the MELIORA-SURVIVORS Study targeting BC survivors (conducted in Lithuania, Spain, Sweden), involving a total of 2,080 participants. The studies will encompass both urban and rural regions and will include participants across the socioeconomic spectrum and/or ethnic minority groups, allowing for the evaluation of how these factors moderate the effectiveness of the MELIORA behavioural change intervention. The studies will follow a randomized-controlled design. For the MELIORA-HEALTHY study, a total of 1080 adult women (360 per site), free of cancer and with at least one behavioural (i.e. low levels of physical activity, unhealthy diet, increased alcohol consumption) or metabolic (i.e. increased BMI) risk factor will be recruited. For the MELIORA-PATIENTS study, a total of 400 adult women diagnosed with BC and currently undergoing treatment (200 per site) will be recruited. For the MELIORA-SURVIVORS study, a total of 600 adult women diagnosed with BC and have completed primary therapy (200 per site) will be recruited.

Participants at each site will be randomly assigned (1:1 allocation) to either the intervention group or the control group. The control group will receive the standard of care that is generic advice for a healthy lifestyle and BC prevention. The intervention group will receive the same generic advice along with the MELIORA VC intervention app. The total study duration for each participant will be 12 months, divided into two six-month periods: the intervention period and the follow-up period. Targeted behaviours will be assessed at three time points: baseline (0 months), end of the six-month intervention period (6 months), and end of the six-month follow-up period (12 months). The primary outcome that will be assessed is physical activity while secondary outcomes include sedentary behaviours, diet, alcohol consumption and health-related quality of life.

The MELIORA project represents an innovative approach to BC prevention by integrating an AI-driven digital health solution into real-world settings. The MELIORA studies highlight the role of technology in promoting sustainable behaviour change to prevent the onset or recurrence of BC. The VC tool that will be developed, tested and evaluated is a key outcome of the MELIORA project and aims to support preventive policies and health promotion guidelines for BC prevention. If successful, the MELIORA VC model could be expanded to other at-risk populations, reinforcing the potential of AI-driven, cost-effective health interventions in cancer prevention. Findings will provide valuable insights for policymakers and healthcare professionals on the feasibility, effectiveness, and cost-effectiveness of AI-supported lifestyle interventions, shaping future public health strategies.

ELIGIBILITY:
Inclusion Criteria:

MELIORA-HEALTHY study participants must meet all of the following criteria in order to be deemed eligible for study participation:

* Reside in Greece, Lithuania, or Spain.
* Be female and at least 18 years of age.
* Have access to and be able to use a smartphone (iOS or Android) compatible with the MELIORA app.
* Be willing and able to use the MELIORA app for the entire study duration.
* Willing to provide informed consent to participate in the study.
* Have at least one of the following behavioural or metabolic risk factors for BC, assessed in a random order (each site may determine the order that is most convenient for them) until eligibility is confirmed. If a risk factor is identified, the subsequent assessments can be skipped:
* Increased alcohol consumption: More than 1 drink per day.
* Increased body mass index (BMI): BMI ≥ 25 kg/m².
* Physical inactivity: Not meeting World Health Organization (WHO) guidelines of at least 150 minutes of moderate-intensity or 75 minutes of high-intensity aerobic exercise per week.
* Suboptimal diet: Low diet quality based on the rapid Prime Diet Quality Score Screener (rPDQS).

MELIORA-PATIENTS study participants must meet all of the following criteria in order to be deemed eligible for study participation:

* Reside in Spain or Lithuania.
* Be female and at least 18 years old.
* Have access to and be able to use a smartphone (iOS or Android) compatible with the MELIORA app.
* Be willing and able to use the MELIORA app for the entire study duration.
* Willing to provide informed consent to participate in the study.
* Have been diagnosed with breast cancer (BC) within the last 6 months and/or currently undergoing treatment (chemotherapy, radiotherapy, immunotherapy, hormone therapy) and/or in active follow-up.

MELIORA-SURVIVORS study participants must meet all of the following criteria in order to be deemed eligible for study participation:

* Reside in Spain, Lithuania, or Sweden.
* Be female and at least 18 years old.
* Have access to and be able to use a smartphone (iOS or Android) compatible with the MELIORA app.
* Be willing and able to use the MELIORA app for the entire study duration.
* Willing to provide informed consent to participate in the study.
* Have completed primary treatment for breast cancer (surgery, chemotherapy, radiotherapy, immunotherapy, targeted therapy, etc.) and currently be in remission.
* Have at least one of the following behavioural or metabolic risk factors for BC, assessed in a random order (each site may determine the order that is most convenient for them) until eligibility is confirmed. If a risk factor is identified, the subsequent assessments can be skipped:
* Increased alcohol consumption: More than 1 drink per day.
* Increased body mass index (BMI): BMI ≥ 25 kg/m².
* Physical inactivity: Not meeting World Health Organization (WHO) guidelines of at least 150 minutes of moderate-intensity or 75 minutes of high-intensity aerobic exercise per week.
* Suboptimal diet: Low diet quality based on the rapid Prime Diet Quality Score Screener (rPDQS).

Exclusion Criteria:

MELIORA-HEALTHY study participants will be excluded from study participation if they meet any of the following criteria:

* Inability to provide fully informed consent.
* Inability to understand or communicate in the local language i.e. Greek in Greece, Lithuanian in Lithuania, Spanish in Spain.
* Current or past diagnosis of cancer or other uncontrolled chronic diseases (e.g., cardiovascular disease, diabetes) that affect lifestyle, dietary habits, or communication skills.
* Mental illness or disorders that affect lifestyle, dietary habits, or communication skills.
* Use of medication that affects lifestyle, dietary habits, or communication skills.
* Recreational drug use.
* Pregnancy, lactation, or intention to become pregnant shortly before, during, or after the intervention.
* Participation in another clinical trial or program aimed at promoting behavioural changes or weight loss at the time of recruitment. If subjects already use health-related apps that affect their weight and lifestyle, including dietary habits and physical activity, the research team will ask them to pause their use until the end of the 12-month study period. However, the use of these applications by the participants cannot be controlled.

MELIORA PATIENTS and MELIORA SURVIVORS study participants will be excluded from study participation if they meet any of the following criteria:

* Inability to provide fully informed consent.
* Inability to understand or communicate in the local language (i.e., Lithuanian in Lithuania, Spanish in Spain, Swedish in Sweden), unless appropriate translation support is available to ensure full understanding of study procedures and informed consent.
* Current or past diagnosis of cancer (other than breast cancer, except skin cancer treated with surgery only) or other uncontrolled chronic diseases (e.g., cardiovascular diseases, diabetes) that affect lifestyle, dietary habits, or communication skills.
* Mental illness or disorders that affect lifestyle, dietary habits, and communication skills.
* Use of medication that affects lifestyle, dietary habits, or communication skills.
* Recreational drug use.
* Pregnancy, lactation, or intention to become pregnant shortly before, during, or after the intervention.
* Participation in another clinical trial or program to promote behavioural changes or weight loss during recruitment. Suppose participants are already using health-related apps affecting their weight and lifestyle, including dietary habits and physical activity. In that case, they will be asked to suspend their use until the end of the 12-month study period. However, the research team cannot control the use of these applications by the participants.
* Severe adherence issues with previous treatments that may interfere with compliance with study tasks (subject to the investigator's assessment).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2080 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Physical activity levels - MVPA minutes | From baseline (T0) until the end of the six-month intervention period (T1)
  The primary outcome will be the mean change in physical activity levels as measured by MVPA minutes from baseline at the end of the six-month intervention period between the intervention and the control group.
Physical activity levels - Step count | From baseline (T0) until the end of the six-month intervention period (T1)
  The primary outcome will be the mean change in physical activity levels as measured by step count from baseline at the end of the six-month intervention period between the intervention and the control group.

SECONDARY OUTCOMES:
Physical activity levels - MVPA minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in physical activity levels as measured by MVPA minutes, from baseline until the end of the 6-month intervention period, within groups.
Physical activity levels - MVPA minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in physical activity levels as measured by MVPA minutes, from baseline until the end of the 6-month follow-up period between groups.
Physical activity levels - MVPA minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in physical activity levels as measured by MVPA minutes, from baseline until the end of the 6-month follow-up period within groups.
Physical activity levels - Step count | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in physical activity levels as measured by step count, from baseline until the end of the 6-month intervention period, within groups.
Physical activity levels - Step count | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in physical activity levels as measured by step count, from baseline until the end of the 6-month follow-up period, between groups.
Physical activity levels - Step count | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in physical activity levels as measured by step count, from baseline until the end of the 6-month follow-up period, within groups.
Aerobic exercise minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in aerobic exercise minutes, from baseline until the end of the 6-month intervention period between groups.
Aerobic exercise minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in aerobic exercise minutes, from baseline until the end of the 6-month intervention period, within groups.
Aerobic exercise minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in aerobic exercise minutes, from baseline until the end of the 6-month follow-up period, between groups.
Aerobic exercise minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in aerobic exercise minutes, from baseline until the end of the 6-month follow-up period, within groups.
Muscle strengthening minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in muscle strengthening minutes, from baseline until the end of the 6-month intervention period within groups.
Muscle strengthening minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in muscle strengthening minutes, from baseline until the end of the 6-month intervention period between groups.
Muscle strengthening minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in muscle strengthening minutes, from baseline until the end of the 6-month follow-up period, within groups.
Muscle strengthening minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in muscle strengthening minutes, from baseline until the end of the 6-month follow-up period, between groups.
Sedentary minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in sedentary minutes, from baseline until the end of the 6-month intervention period between groups.
Sedentary minutes | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in sedentary minutes, from baseline until the end of the 6-month intervention period within groups.
Sedentary minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in sedentary minutes, from baseline until the end of the 6-month follow-up period, within groups.
Sedentary minutes | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in sedentary minutes, from baseline until the end of the 6-month follow-up period, between groups.
Αlcohol consumption | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in alcohol consumption (servings/week), from baseline until the end of the 6-month intervention period within groups.
Αlcohol consumption | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in alcohol consumption (servings/week), from baseline until the end of the 6-month intervention period between groups.
Αlcohol consumption | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in alcohol consumption (servings/week), from baseline until the end of the 6-month follow-up period, within groups.
Αlcohol consumption | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in alcohol consumption (servings/week), from baseline until the end of the 6-month follow-up period, between groups.
Diet quality | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in rapid Prime Diet Quality Score Screener (rPDQS) diet score (0-26 points with higher scores meaning a better diet quality) and individual dietary components, from baseline until the end of the 6-month intervention period within groups.
Diet quality | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in rapid Prime Diet Quality Score Screener (rPDQS) diet score (0-26 points with higher scores meaning a better diet quality) and individual dietary components, from baseline until the end of the 6-month intervention period between groups.
Diet quality | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in rapid Prime Diet Quality Score Screener (rPDQS) diet score (0-26 points with higher scores meaning a better diet quality) and individual dietary components, from baseline until the end of the 6-month follow-up period, within groups.
Diet quality | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in diet score and individual dietary components, from baseline until the end of the 6-month follow-up period, between groups.
Health-related quality of life | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in quality of life [EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L, scale 1-5 with greatest values meaning worst outcomes)] , from baseline until the end of the 6-month intervention period within groups.
Health-related quality of life | From Baseline (T0) until the end of the six-month intervention period (T1)
  Mean changes in quality of life [EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L, scale 1-5 with greatest values meaning worst outcomes)], from baseline until the end of the 6-month intervention period between groups.
Health-related quality of life | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in quality of life [EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L, scale 1-5 with greatest values meaning worst outcomes)], from baseline until the end of the 6-month follow-up period, within groups.
Health-related quality of life | From Baseline (T0) until the end of the 6-month follow-up period (T2)
  Mean changes in quality of life [EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L, scale 1-5 with greatest values meaning worst outcomes)], from baseline until the end of the 6-month follow-up period between groups.

OTHER OUTCOMES:
Body mass index (BMI) | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in BMI, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups.
Role modelling behaviours | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in role modelling behaviours, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. An eleven-item tool was developed specifically for the purpose of this research to assess the potential impact of the intervention on health behaviours of participants' daughters. These items assess mothers' efforts to inform their daughter(s) about their participation in the intervention, to practise health behaviours in front of or along with their daughter(s), and to motivate their daughter(s) to also improve their health behaviours, as well as the perceived effect of mothers' participation on the daughter(s)' eating habits, physical activity, sedentary behaviour, alcohol consumption, and health literacy.
Health literacy | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in health (European Health Literacy Survey Questionnaire (HLS-EU-Q) using 4-point Likert scales ranging from 1 = very easy to 4 = very difficult) from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups.
e-health literacy | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in e-health literacy (modified version of the Application subscale of the eHealth Literacy Scale in Web 3.0 context (eHLS Web 3.0) that uses 5-point Likert scales ranging from 1 = strongly disagree to 5 = strongly agree) from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups.
Psychosocial parameters - Physical capability | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in physical capability, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. Physical capability will be measured with a modified version of the physical competence subscales of the Physical Literacy in Adults Scale (PLAS), which assess one's perceived physical strength (3 items) and coordination/ balance (3 items) using 7-point Likert scales ranging from 1 = very untrue to 7 = very true.
Psychosocial parameters - Psychological capability | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in psychological capability, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. A 6-item scale developed by Sniehotta, Scholz, & Schwarzer (2005) and later adapted by Willmott, Pang, & Rundle-Thiele (2021) will be used to assess the extent to which participants tried to self-monitor their physical activity behaviour (i.e., action control) in the last four weeks using 7-point Likert scales ranging from 1 = very untrue to 7 = very true.
Psychosocial parameters - Psychological capability | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in psychological capability, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. A10-item scale (Sniehotta, Schwarzer, Scholz, & Schüz, 2005) will be employed to assess the extent to which participants have planned when, where, how often, and how to engage in physical activity (i.e., action planning, 4 items) as well as how to overcome potential barriers for being physically active (i.e., coping planning, 6 items) using 4-point Likert scales ranging from 1 = completely disagree to 4 = totally agree.
Psychosocial parameters - Social support for physical activity | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in social support for physical activity, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. Social support for physical activity will be measured with the Exercising together subscale (5 items) of the Social Support for Exercise Behaviour Scale (SSEBS) (Sallis, Grossman, Pinski, Patterson, & Nader, 1987), as used in Howlett, Schulz, Trivedi, Troop, & Chater (2019). Specifically, participants will indicate how often their friends and family members supported them in being physically active during the past three months using 5-point Likert scales ranging from 1 = none to 5 = very often.
Psychosocial parameters - Reflective motivation | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in reflective motovation, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. The 5-item self-efficacy for physical activity scale by Marcus, Selby, Niaura, & Rossi (1992) will be used to assess participants' confidence in their ability to perform physical activity under various challenging circumstances. The measurement instrument uses 5-point Likert scales ranging from 1 = not confident at all to 5 = extremely confident and has been extensively used in prior research to assess self-efficacy for physical activity.
Psychosocial parameters - Automatic motoivation | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in automatic motivation, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. The International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) (Thomson, 2007) will be used to assess positive (5 items) and negative (5 items) affective responses towards physical activity, as used in Willmott, Pang, & Rundle-Thiele (2021). The measurement instrument uses 5-point Likert scales ranging from 1 = never to 5 = always to assess to what extent an individual generally feels positive and negative emotions about physical activity.
Psychosocial parameters - Injunctive social norms for physical activity | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in injunctive social norms for physical activity, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. Injunctive social norms for physical activity will be assessed with two items developed by Courneya, Friedenreich, Arthur, & Bobick (1999), which measure the extent to which important others expect or support the individual to be physically active in the coming 4 months.
Psychosocial parameters - Descriptive norms for physical activity | From Baseline (T0) until the end of the six-month intervention period (T1) and from T0 until the end of the 6-month follow-up period (T2)
  Mean changes in descriptive norms for physical activity, from baseline until the end of the 6-month intervention period and until the end of the 6-month follow-up period, within and between groups. Descriptive norms will be assessed with three items, measuring to what extent family, friends, and co-workers engage in physical activity themselves (Rhodes & Courneya, 2003). Both measurement instruments use 7-point Likert scales ranging from 1 = strongly disagree to 7 = strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Professor, Principal Investigator — Department of Nutrition and Dietetics, School of Health Science & Education, Harokopio University, Athens, Greece
Locations (7):
- Harokopio University, Athens, Greece
- Lithuania (2):
  - Lietuvos Sveikatos Mokslų Universitetas (Lsmu), Kaunas
  - Pagalbos Onkologiniams Ligoniams Asociacija (Pola L T), Kaunas
- Spain (2):
  - Fundación Para El Fomento de La Investigación Sanitaria Y Biomédica de La Comunitat Valenciana (Fisabio), Valencia
  - INCLIVA - Instituto de Investigación Sanitaria, Valencia
- Sweden (2):
  - Bröstcancerföreningen Amazona I Stockholms Län (Amazona), Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: MELIORA website link — https://melioraproject.eu/